CLINICAL TRIAL: NCT07299643
Title: The Application of 3DSlicer Technology in Percutaneous Nephrolithotomy Surgery.
Brief Title: Application of 3DSlicer Technology in Percutaneous Nephrolithotomy Surgery.
Status: Completed | Type: Observational
Sponsor: Ting Huang (Other)
Responsible Party: Sponsor-Investigator, Ting Huang, Principal Investigator, Zhejiang University
Organization: Zhejiang University (Other)
Other Study IDs: 2022282
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Percutaneous Nephrolithotomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stone Free Group
- Stone Residue Group

SUMMARY:
Objectives: Percutaneous nephrolithotomy (PCNL) has become a widely used technique for managing renal calculi. However, the rate of residual stones remains high. Accurate preoperative assessment of the individual's renal collecting system anatomy and strategic planning of access pathways are essential for improving stone-free outcomes. This study investigated whether characteristics of the target calyx can predict stone clearance through a distinct puncture calyx and developed a model to estimate the risk of residual stones in the target calyx.

Methods: We performed a retrospective analysis of patients who underwent PCNL in the urology department of our center between January 2023 and June 2025, in whom the puncture calyx differed from the target calyx (67 cases with complete stone clearance and 38 cases with residual stones). Three-dimensional reconstructions of the renal collecting system and calculi were generated from preoperative urinary tract CT scans, and spatial parameters were obtained from these models. Patient and stone characteristics were combined with 3D-derived variables for binary logistic regression to identify predictive factors and construct nomograms. Model performance was assessed using receiver operating characteristic (ROC) and calibration curves, while clinical utility was evaluated through decision curve analysis (DCA). The Youden index was applied to determine the optimal cutoff value.

ELIGIBILITY:
Inclusion Criteria:

① preoperative diagnosis of renal calculi confirmed by computed tomography urography (CTU); ② completion of standard-channel (F24) PCNL with the puncture and target calyces situated in different renal calyces; and ③ postoperative CT imaging performed within one week after surgery.

Exclusion Criteria:

① anatomical abnormalities of the affected kidney, such as severe renal rotation or horseshoe kidney; and ② history of secondary procedures, including repeat PCNL or renal puncture with fistula formation.

Ages: 28 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: After applying these criteria, a total of 105 renal calyces were included for analysis
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
predict the stone free possibility of kidey stone | 2023-2025
  AUC curve
predict the stone free possibility of kidey stone | 2023-2025
  DCA curve

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Affiliated Jinhua Hospital, Zhejiang University School of Medicine,, Jinhua, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No